CLINICAL TRIAL: NCT03166046
Title: Migraine Prevention Using Pulsed Shortwave Therapy
Brief Title: Migraine Prevention Using ActiPatch
Acronym: PSWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAIRB-17-0021
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled trial using an active pulsed shortwave therapy device or placebo pulsed shortwave therapy device
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Coded devices that are identical in appearance and function. Placebo device does not emit electromagnetic field. Active device electromagnetic field is sub-sensory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study Group (Active Comparator): Subjects will use the active pulsed shortwave therapy device (ActiPatch) as a prophylactic treatment for episodic migraine
  Interventions: Device: Pulsed Shortwave Therapy
- Control Group (Placebo Comparator): Subjects will use the placebo pulsed shortwave therapy device (Placebo ActiPatch) as a prophylactic treatment for episodic migraine
  Interventions: Device: Placebo Pulsed Shortwave therapy

INTERVENTIONS:
Device: Pulsed Shortwave Therapy — Stimulation of the supratrochlear and supraorbital branches of the ophthalmic nerve.
  Other Names: ActiPatch
  Arms: Study Group
Device: Placebo Pulsed Shortwave therapy — Placebo Stimulation of the supratrochlear and supraorbital branches of the ophthalmic nerve.
  Other Names: Placebo ActiPatch
  Arms: Control Group

SUMMARY:
Chronic pain is now widely understood to be due to central sensitization, which leads to exaggerated pain perception. Migraine is no exception, since it is well known that sensitization of the trigeminovascular pain pathway can occur during a migraine attach. There is early evidence that ActiPatch can help mitigate this sensitization, so this study is being conducted to determine the efficacy of ActiPatch in preventing chronic, episodic migraines.

DETAILED DESCRIPTION:
Migraine is a common neurological disorder characterized by episodes of unilateral or bilateral headache lasting for hours to days, which may be accompanied by photophobia, phonophobia, nausea and vomiting. Pharmacological management is the first treatment option for subjects with migraine. However, some patients do not tolerate acute and/or prophylactic medicine due to side effects or contraindications due to comorbidity of other diseases or due to a wish to avoid medication for other reasons. The risk of medication overuse due to frequent migraine attacks represents a major health hazard with direct and indirect cost concerns. The prevalence of medication overuse headache is 1 -2% in the general population, that is, about half the population suffering chronic headache (15 headache days or more per month) have medication overuse headache.It is well-known that a primary brain dysfunction leads to episodic activation and sensitization of the trigeminovascular pain pathway during attacks. However, a functional and anatomic relationship exists between peripheral afferent nerves supplying the head and neck and the brainstem, subcortical and higher order brain processing centers. There is some evidence that interventions targeting peripheral nerves are able to modulate neuronal circuits involved in pain control and that they could be useful in some selected patients with migraine.

Supraorbital neurostimulation (tSNS) of the upper branches of the trigeminal nerves was found superior to sham stimulation for episodic migraine prevention in a previous randomized trial in a large cohort of patients with migraine. In this study the pulsed shortwave device will be incorporated in a wrap which will enable easy placement of the device in the desired located which will be over the supratrochlear and supraorbital branches of the ophthalmic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Male or female ages 18 or above with migraine headache
* 3 or greater occurrences of migraine per month
* no prior use of neuromodulation for migraine headache

Exclusion Criteria:

* Female participant who is pregnant
* prior use of neuromodulation for migraine headache
* Laminectomy, laminotomy or discectomy within 12 months of enrollment.
* Active psychiatric disorders will be excluded (e.g. use of antipsychotic medication, bipolar disorder, schizophrenia).
* Patients diagnosed with history of significant mood disorder will be excluded (e.g., depression or anxiety with adequate control would be acceptable).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Migraine frequency | 4 weeks
  frequency of migraine attacks
Migraine duration | 4 weeks
  Duration of migraine attacks

SECONDARY OUTCOMES:
Migraine intensity measured with Visual Analogue Pain Score | 4 weeks
  Migraine intensity measured with visual analogue pain score (VAS scores)
Headache disability measured with Headache Impact Test | 4 weeks
  Headache impact test (HIT-6)

CONTACTS AND LOCATIONS:
Overall Officials: Sree Koneru, Ph.D., Study Director — BioElectronics Corporation; Barry Eppley, MD, Principal Investigator — Eppley Group; Ian Rawe, Ph.D., Study Chair — BioElectronics Corporation
Locations (1):
- Eppley Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No